CLINICAL TRIAL: NCT00822107
Title: A Translational Approach to Gitelman Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Oregon Clinical and Translational Research Institute (Other)
Responsible Party: Principal Investigator, David Ellison, Professor of Medicine, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00004529
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Gitelman Syndrome
Keywords: Hypokalemia; Bartter Syndrome; Salt Wasting
MeSH Terms: conditions — Gitelman Syndrome; Hypokalemia; Bartter Syndrome | interventions — Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thiazide Response (Experimental): Hydrochlorothiazide 50 mg will be administered by mouth once.
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Hydrochlorothiazide — 50 mg one time
  Other Names: HCTZ

SUMMARY:
This study will test the response to a single dose of thiazide diuretic as a diagnostic test for Gitelman syndrome. Individuals with hypokalemic alkalosis will be enrolled. After a baseline study, they will have the response to 50 mg hydrochlorothiazide on fractional chloride excretion examined.

DETAILED DESCRIPTION:
The purpose of this study is to test the hypothesis that Gitelman syndrome (GS) can be diagnosed using a simple clinical protocol. GS is an inherited kidney disease that usually shows up in patients as low blood potassium levels. Currently, no commercial genetic test for GS exists. Currently, GS is diagnosed based upon clinical findings but this method is not precise and often not reliable. Thus, in order to develop new treatments specific for GS patients, a more exact method of diagnosis would be of benefit.

Eligible subjects are men and women ages 21-60 with normal blood pressure who have been diagnosed with low blood potassium of uncertain cause. Subjects may withdraw at any time.

This study requires 3 visits to OHSU's campus. Study Visit 1 will occur during a normal visit with the nephrologist. As part of the normal visit, a complete interview, physical exam and urine and blood samples will be taken. In addition, another blood sample will be taken and used for genetic analysis. A urine pregnancy test will be administered. A Quality of Life survey, described below, will be administered. The genetic analysis, urine pregnancy test and Quality of Life survey are not normal tests for GS. Blood and urine samples, as well as pregnancy tests will be collected/administered at the Oregon Clinical and Translational Research Institute (OCTRI).

During the intervention period, subjects will refrain from taking their potassium sparing medications for 7 days. This period is called the washout period and is needed to ensure that blood tests during the hydrochlorthiazide (HCTZ, a "water pill") (see below), are not affected by medications. On the 3rd day of the washout period, Study Visit 2 will occur at the OCTRI. This will require blood to be drawn, to insure that subjects maintain proper blood levels of potassium and magnesium. Magnesium and potassium supplements will be allowed during the washout. After review of the blood test results, the investigator may adjust the doses of these supplements in order to keep subject blood levels of potassium and magnesium as close to normal as possible. Blood pressure, heart rate and breathing rate will also be checked at this visit.

Study Visit 3 will occur at the OCTRI and will be devoted to the HCTZ test. During the course of the HCTZ test, subjects will have an plastic tube (an IV) placed in an arm vein, have vital signs checked and receive 50mg of HCTZ to take by mouth . Subjects will provide 8 urine samples and 3 blood samples. The time required for this visit is expected to be 6 hours.

The total time required for subjects to complete the study from Study Visit 1 through discharge from the OCTRI on Study Visit 3 will not be less than 9 days and subjects should not expect the total length to exceed three weeks depending on available appointments for Study Visit 3 at the OCTRI.

The Quality of Life survey is derived from a national research corporation and has been modified for use in this study. The authors of this survey allow free public use of this document provided it is properly referenced in any presentation of the study's results.

HCTZ is an FDA approved medication. There are no experimental drugs or devices used in this study.

The purpose of this study is to develop methods for, and determine the feasibility of, performing a HCTZ test and genetic analysis for GS at OHSU. There is no statistical analysis of data, but descriptive characteristics will be entered into an Access database with password restricted access. Genetic samples will be analyzed using PCR and standard sequencing techniques. Data and samples will be stored for a maximum of 15 years.

ELIGIBILITY:
Inclusion Criteria:

1. Institutional Review Board (IRB) approved written Informed Consent and Health Insurance Portability and Accountability Act (HIPAA) Authorization as per national regulations, must be obtained from the subject or legally authorized representative prior to any study-related procedures (including withdrawal of prohibited medication, if applicable).
2. Subject is between the ages of 21 and 60.
3. Female subjects of child bearing potential must have a negative urine pregnancy test at the screening visit (Study Visit 1) and must agree to maintain effective birth control during the study.
4. Subjects who are referred to Dr. Ellison for evaluation of normotensive hypokalemia of unknown etiology

Exclusion Criteria:

1. Subject has known allergy to thiazide or sulfonamide medications
2. Subject is pregnant or lactating.
3. Subject has major systemic illnesses that affect potassium regulation through pathology or pharmacologic treatment. This category includes:

   * Hypertension
   * Requiring regular pharmacological control
   * History of blood pressure greater than 140mmHg systolic and 90mmHg diastolic
   * Congestive heart failure
   * Cirrhosis of the liver
4. Subject has documented kidney disease resulting in anuria, proteinuria or abnormal urinalysis, or requiring dialysis for treatment.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Ellison, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thiazide Response
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Thiazide Response
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 42 [38 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Chloriuretic Response to a Thiaizde
Description: Change from baseline in fractional chloride excretion in response to a single dose of hydrochlorothiazide
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: fractional chloride excretion
Arm/Group | Thiazide Response
Number analyzed (Participants) | 5
fractional chloride excretion | 1.23 (0.93)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Thiazide Response
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No